CLINICAL TRIAL: NCT07213791
Title: A Dose Escalation and Dose Optimization Phase 1a/1b Study to Evaluate Safety, Tolerability and Dosimetry of Radioligand Therapy With LY4337713 in Adults With FAP-Positive Solid Tumors (FiREBOLT)
Brief Title: A Study of LY4337713 in Participants With FAP-Positive Solid Tumors
Acronym: FiREBOLT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 27513; J6K-OX-JSFA (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-10-07; First posted 2025-10-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Neoplasms; Breast Neoplasms; Pancreatic Intraductal Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Cholangiocarcinoma
Keywords: Cancer-associated fibroblasts (CAF); Lutetium-177; LuFAP; Lu-177-FAP
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Pancreatic Intraductal Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY4337713 (Cohort A1) (Experimental): Escalating doses of LY4337713 administered intravenously (IV).
  Interventions: Drug: LY4337713
- LY4337713 (Cohort A2) (Experimental): Two or more dose regimens of LY4337713 (evaluated during dose escalation) administered IV.
  Interventions: Drug: LY4337713
- Experimental: LY4337713 (Cohort B) (Experimental): Tumor specific cohort will receive LY4337713 administered IV.
  Interventions: Drug: LY4337713
- Experimental LY4337713 (Cohort C) (Experimental): Tumor specific cohort will receive LY4337713 administered IV.
  Interventions: Drug: LY4337713
- Experimental: LY4337713 (Cohort D) (Experimental): Tumor specific cohort will receive LY4337713 administered IV.
  Interventions: Drug: LY4337713
- LY4337713 (Cohort E) (Experimental): Tumor specific cohort will receive LY4337713 administered IV.
  Interventions: Drug: LY4337713

INTERVENTIONS:
Drug: LY4337713 — Administered IV.

SUMMARY:
This is a study of LY4337713 in participants with certain types of cancer that is advanced or has spread. Participants must have cancer with high levels of a protein called fibroblast activation protein (FAP). The purpose of this study is to evaluate safety, side effects, and efficacy of LY4337713. In addition, this study will evaluate how much LY4337713 gets into the bloodstream, how it is broken down, and how long it takes the body to get rid of it. For each participant, the study will last about 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Must have clinical or imaging evidence of fibroblast activation protein (FAP) expression per local assessment
* Must have histologically or cytologically confirmed diagnosis of one of the following:

  * Adenocarcinoma of the pancreas
  * Hormone receptor (HR)-positive human epidermal growth factor 2 (HER2)-negative breast cancer
  * HER2-positive breast cancer
  * Triple negative breast cancer (TNBC)
  * Platinum-resistant or refractory ovarian cancer
  * Other solid tumors

    * Gastric cancer (adenocarcinoma)
    * Colorectal cancer (CRC)
    * Esophageal cancer (squamous cell carcinoma or adenocarcinoma)
    * Cholangiocarcinoma
* Must have received prior treatments as indicated below:

  * Phase 1a

    * Adenocarcinoma of the pancreas: Participants must have progressed after at least 1, but no more than 2 prior regimens for locally advanced unresectable or metastatic disease.
    * HR-positive HER2-negative breast cancer: Participants must have received less than or equal to (≤)5 prior lines of treatment for advanced or metastatic disease, which must include a cyclin-dependent kinase 4/6 inhibitor.
    * HER2-positive breast cancer: Participants must have progressed on at least 2 lines of HER2-targeted therapy, which should include at least 1 antibody-drug conjugate (ADC) for metastatic disease (if locally available).
    * TNBC: Participants must have progressed on at least 2 lines of therapy for metastatic disease.
    * Platinum-resistant or refractory ovarian cancer: Participants must have progressed on or after at least 1 platinum-based therapy.
    * Other solid tumors (gastric cancer, CRC, esophageal and cholangiocarcinoma): Participants must have received greater than or equal to (≥)1 prior line of systemic therapy for advanced or metastatic disease; including prior line(s) in combination with immunotherapy or vascular endothelial growth factor inhibitor.
  * Phase 1b:

    * Participants must have advanced or metastatic solid tumors and have received ≥1 prior line of therapy.
* Must have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1.
* Measured creatinine clearance ≥60 milliliters per minute (mL/min)

Exclusion Criteria:

* Have known active central nervous system (CNS) metastases or carcinomatous meningitis.
* Have history of Grade 4 myelosuppression lasting greater than (>)7 days, or Grade 3 myelosuppression requiring more than 6 weeks recovery.
* Have significant cardiovascular disease
* Have prolongation of the corrected QTcF >470 milliseconds (msec) during screening. QTcF is calculated using Fridericia's Formula: QTcF = QT/(RR0.33)
* Have evidence of ongoing and untreated urinary tract obstruction
* Had previous hemi- or total-body radiation.
* Had previous adoptive T-cell therapy (e.g., chimeric antigen receptor T-cell [CAR-T therapy, T-cell receptor [TCR] therapy, etc.)
* Unable to lie flat during, or otherwise tolerate, single photon emission computed tomography (SPECT), positron emission tomography (PET), computed tomography (CT) or magnetic resonance imaging (MRI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Percentage of Participants with Dose Limited Toxicity (DLT) Toxicities | Cycle 1 (28 days)
Phase 1b: Objective Response Rate (ORR): Percentage of Participants with Best Response of Complete Response (CR) or Partial Response (PR) | Baseline through imaging follow-up, up to 5 years
  Per investigator assessed Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
Phase 1a: Absorbed Dose Estimates (Gy) in Normal Organs | Baseline through Cycle 4 Day 4 (Cycle = 4 or 6 weeks)
Phase 1a: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY4337713 | Cycle 1 Day 1 up to Cycle 2 Day 4 post dose (Cycle = 4 or 6 weeks)
Phase 1a: PK: Area Under the Concentration Time Curve (AUC) of LY4337713 | Cycle 1 Day 1 up to Cycle 2 Day 4 post dose (Cycle = 4 or 6 weeks)
Phase 1a: Objective Response Rate (ORR): Percentage of Participants with Best Response of Complete Response (CR) or Partial Response (PR) | Baseline through imaging follow-up, up to 1 year
  Per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Phase 1a: Number of Participants with Best Overall Response (BOR) | Baseline through imaging follow-up, up to 1 year
  Best response recorded from the start of study treatment until the earliest of objective disease progression or start of new anticancer therapy, per RECIST v1.1.
Phase 1a and 1b: Duration of Response (DOR) | Baseline through imaging follow-up, up to 5 years
  Time between the date of first documented response of CR or PR to the date of first disease progression, as assessed by the investigator per RECIST v1.1 or death due to any cause, whichever occurs first.
Phase 1a and 1b: Time to Response (TTR) | Baseline through imaging follow-up, up to 1 year
  Time from first dose date to the date of first documented response of CR or PR
Phase 1a and 1b: Percentage of Participants with Disease Control Rate (DCR) | Baseline through imaging follow-up, up to 1 year
  Percentage participants who achieved a BOR of CR, PR, or stable disease (SD), per RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- United States (18):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford University Medical Center, Stanford, California
  - Biogenix Molecular, LLC, Miami, Florida
  - Indiana University (IU) School of Medicine, Indianapolis, Indiana
  - United Theranostics, Glen Burnie, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - BAMF Health Inc., Grand Rapids, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - New York University (NYU) Clinical Cancer Center, New York, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Texas Oncology - DFW (Sammons CC), Dallas, Texas
  - University of Wisconsin - Carbone Cancer Center, Madison, Wisconsin
- Universitaetsklinikum Essen, Essen, Germany
- Netherlands (6):
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek Ziekenhuis (NKI-AVL), Amsterdam
  - Amsterdam UMC - Locatie VUmc, Amsterdam
  - Erasmus MC, GE Rotterdam
  - Maastricht University Medical Center, Maastricht
  - Stichting Radboud Universitair Medisch Centrum, Nijmegen
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to Lilly Trials — https://trials.lilly.com/en-US/trial/660077